CLINICAL TRIAL: NCT01531790
Title: A Phase I Study of Continuous Endostar Intravenous Infusion Combined With Pemetrexed and Carboplatin in Advanced NSCLC Patients
Brief Title: A Study of Continuous Endostar Intravenous Infusion Combined With Pemetrexed and Carboplatin in Advanced Non Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-93
Record Dates: First submitted 2012-02-07; First posted 2012-02-13 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Endostar; Carboplatin; Pemetrexed; NSCLC; Phase I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endostar plus pemetrexed/carboplatin (Experimental): 21 days as one cycle, for a total of 4-6 cycles
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Endostar; Drug: Centrum

INTERVENTIONS:
Drug: Carboplatin — d1, AUC 5, i.v.
Drug: Pemetrexed — d1, 500 mg/m2, i.v.
Drug: Endostar — d2-d21, continuous Endostar intravenous infusion, 7.5 mg/m2/d, 15 mg/m2/d or 30 mg/m2/d, etc.
Drug: Centrum — 1 tablet/day

SUMMARY:
This study is to evaluate the safety, tolerability, clinical efficacy and pharmacokinetics of continuous Endostar intravenous infusion combined with pemetrexed and carboplatin in advanced non small cell lung cancer (NSCLC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of inoperable stage IIIB/IV non-squamous NSCLC
* At least one measurable lesion (RECIST criteria)
* Life expectancy > 3 months
* ECOG performance status 0-2
* Adequate hematologic function: WBC ≥ 3.0×109 /L，ANC ≥ 1.5×109 /L，Hb ≥ 90 g/L，PLT ≥ 100×109 /L
* Adequate renal, hepatic and coagulation function
* Written informed consent

Exclusion Criteria:

* With uncontrollable malignant pleural effusion or ascites
* Thoracic or abdominal surgery within 28 days prior to study entry
* History of cerebral stroke or TIA within 6 months prior to study entry
* With uncontrollable hypertension, hypertensive emergency or hypertensive encephalopathy
* Arrhythmia in need of antiarrhythmic treatment, history of angina pectoris, myocardial infarction, myocardial ischemia or congestive heart failure (> NYHA class II)
* With serious infection (> NCI CTC grade 2)
* Gastrointestinal perforation, fistula formation, and/or intra-abdominal abscess within 6 months prior to study entry
* Symptomatic brain metastases
* Patient who has epilepsy
* History of HIV infection or chronic hepatitis B or C
* Allergic to any of the study drugs
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | up to 21 days

SECONDARY OUTCOMES:
Objective Response Rate | up to 6 cycles
Disease Control Rate | up to 6 cycles
Progression-free Survival | up to 2 years
Overall Survival | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China